CLINICAL TRIAL: NCT05518825
Title: Assessment of ONS-flavour Preference in Cancer Patients With and Without Taste Alterations
Acronym: PREFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SBB21R&36579
Record Dates: First submitted 2022-08-10; First posted 2022-08-29 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Oncology; Taste, Altered
Keywords: Oral nutritional supplement; Oncology; Taste alterations
MeSH Terms: conditions — Neoplasms; Dysgeusia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fortimel/Nutridrink Compact Protein (Experimental): Twice daily serving of the study product
  Interventions: Dietary Supplement: Fortimel/Nutridrink Compact Protein

INTERVENTIONS:
Dietary Supplement: Fortimel/Nutridrink Compact Protein — Twice daily serving of the study product

SUMMARY:
A single arm intervention study examining ONS-flavour preference in cancer patients with and without taste alterations

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with cancer
2. Undergoing, or having undergone systemic anti-cancer treatment or radiotherapy in the past 12 months.
3. Age > 18 years
4. Written informed consent

Exclusion Criteria:

1. Taste and smell alterations not caused by the cancer or anti-cancer treatment
2. Galactosaemia
3. Use of thickener to be able to swallow safely
4. Allergies to any of the product ingredients or any of the flavours
5. Current prescription for ONS, enteral nutrition or parenteral nutrition
6. Diabetes mellitus Type I or Type II
7. Open sores or severe inflammation in the mouth or throat
8. Undergoing dialysis
9. Hepatic encephalopathy
10. Patients with heart failure who have symptoms of heart failure at rest and/or are unable to carry on any physical activity without discomfort
11. Known pregnancy or lactation
12. Average alcohol use of > 21 glasses per week for men or > 14 glasses per week for women or drug abuse in opinion of the investigator
13. Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
14. Participation in any other studies involving food products concomitantly or within two weeks prior to entry into the study.
15. Employees of Nutricia Research and/or partners, parents, children and brothers/sisters of employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Choice for the Fortimel/Nutridrink Compact Protein sensation flavour over the Fortimel/Nutridrink Compact Protein regular flavour | On 4 days
  Subjects take one sensation flavour and one regular flavour and are asked in a direct question which flavour they prefer.

SECONDARY OUTCOMES:
Difference between average liking scores [score 0-10] for Fortimel/Nutridrink Compact Protein sensation flavour range versus Fortimel/Nutridrink Compact Protein regular flavour range | On 4 days
Choice for the Fortimel/Nutridrink Compact Protein sensation flavours over the Fortimel/Nutridrink Compact Protein regular flavours between patients with and patients without Taste and Smell Alterations | On 4 days
  Subjects take one sensation flavour and one regular flavour and are asked in a direct question which flavour they prefer.
Difference in average liking scores [score 0-10] for Fortimel/Nutridrink Compact Protein sensation flavour versus Fortimel/Nutridrink Compact Protein regular flavour between patients with and patients without Taste and Smell Alterations | On 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nutricia Clinical Research Unit, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No